CLINICAL TRIAL: NCT07322666
Title: Tissue Repair of Incisions for Biopsy and Mouth Ulcers Using Non-Thermal Plasma
Brief Title: Non-Thermal Plasma vs. Low-Level Laser Therapy for Recurrent Oral Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Nuclear Research - Mexico (Other)
Collaborators: Autonomous University of the State of Mexico (Unknown)
Responsible Party: Principal Investigator, Benjamín Gonzalo Rodríguez Méndez, Professional B, Level 19, National Institute of Nuclear Research - Mexico
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEICIEAO-2018-001
Record Dates: First submitted 2025-12-15; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Stomatitis; Aphthous Ulcer
Keywords: Oral Ulcers; Non-Thermal Plasma; Low-Level Laser Therapy; Placebo; Healing; Pain
MeSH Terms: conditions — Stomatitis; Stomatitis, Aphthous; Oral Ulcer; Pain | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment with Non-Thermal Plasma (NTP) (Experimental)
  Interventions: Device: Non-Thermal Plasma (NTP)
- Treatment with Low-Level Laser Therapy (LLLT) (Active Comparator)
  Interventions: Device: Low-Level Laser Therapy (LLLT)
- Treatment with Placebo (Placebo Comparator)
  Interventions: Procedure: Placebo

INTERVENTIONS:
Device: Non-Thermal Plasma (NTP) — Topical application of cold (non-thermal) plasma to the oral ulcer using a plasma generator, with specific time and power parameters.
  Arms: Treatment with Non-Thermal Plasma (NTP)
Device: Low-Level Laser Therapy (LLLT) — Topical application of low-power laser radiation (low-level laser therapy) to the oral ulcer, following a standardized time and wavelength protocol.
  Arms: Treatment with Low-Level Laser Therapy (LLLT)
Procedure: Placebo — Simulation of the application procedure (e.g., turning on a device without active plasma or laser emission, or application with the device turned off) to mask group assignment.
  Arms: Treatment with Placebo

SUMMARY:
The goal of this clinical trial (pilot study) is to evaluate the feasibility and preliminary effectiveness of Non-Thermal Plasma (NTP) in treating pain and accelerating healing in 50 patients with Recurrent Oral Ulcers (ROUs). The main questions it aims to answer are:

Is the study design feasible for a future large-scale trial?

Does NTP show promising preliminary results in reducing ulcer size and healing time compared to standard laser therapy and placebo?

Does NTP provide superior pain relief compared to standard laser therapy and placebo?

Researchers will compare the NTP group (n=20) to the Low-Level Laser Therapy (LLLT) group (n=20) and the placebo group (n=10) to see if NTP is more effective in accelerating healing and reducing pain.

Participants will:

Be randomly assigned to one of three treatment groups (NTP, LLLT, or placebo).

Receive their assigned treatment for their oral ulcers.

Undergo measurements of their ulcer size, report their pain perception using a visual analog scale (VAS), and have their time to complete healing recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age
* Patients of both sexes
* Patients with recurrent oral ulcers (ROU)
* Patients without oral soft tissue diseases
* Patients with at least one recurrent ulcer

Exclusion Criteria:

* Patients under 18 years of age
* Patients with ROU of more than 48 hours' duration
* Patients with gingivitis and/or periodontitis
* Patients undergoing maxillofacial orthopedic and/or orthodontic treatment
* Patients with ill-fitting dentures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-02-04 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Feasibility - Patient recruitment rate | From the start of enrollment to the end of the recruitment period, an average of 1 month.
  Proportion of the target sample size successfully recruited within the recruitment period. Unit of Measure: Percentage (%)
Feasibility - Patient adherence to the intervention protocol | From the first intervention to the last planned session for each participant.
  Proportion of prescribed treatment sessions completed by enrolled participants. Unit of Measure: Percentage (%)
Preliminary efficacy - Time to complete ulcer re-epithelialization | From baseline (day of intervention) until complete healing, assessed daily up to 30 days.
  Number of days required for the ulcer to achieve complete re-epithelialization (visual absence of ulcer crater) confirmed by clinical examination. Unit of Measure: Days
Preliminary efficacy - Change in pain intensity measured by a Visual Analogue Scale (VAS) | From baseline (pre-intervention) to 48 hours post-intervention
  The Visual Analogue Scale (VAS) is a 0 to 10 scale, where "0" represents "no pain" and "10" represents "the worst pain". A higher score indicates worse pain. The change score (post-intervention minus baseline) will be calculated. Unit of Measure: 0-10 VAS

SECONDARY OUTCOMES:
Change in ulcer surface area | From baseline (day of intervention) to days 1, 2, 3, 5, and 7 post-intervention
  Ulcer size will be measured by calculating the surface area from perpendicular diameters (length and width in millimeters) using a standard periodontal probe or digital caliper. Unit of Measure: Square millimeters (mm²)
Safety - Incidence and severity of treatment-related adverse events | From the first intervention until the end of the follow-up period (up to 7 days post-intervention)
  All adverse events and local reactions (e.g., erythema, edema, pain exacerbation) will be recorded and graded for severity using the Common Terminology Criteria for Adverse Events (CTCAE) v5.0 or a similar standardized scale. The relationship to the intervention will be assessed. Unit of Measure: Number of participants with adverse events, and severity grade.
Cumulative use of rescue analgesic medication | From baseline to complete healing or up to 30 days, whichever comes first
  The total amount of rescue analgesic medication (e.g., acetaminophen/paracetamol) consumed by each participant, recorded in a daily diary. Unit of Measure: Milligrams (mg) of medication

CONTACTS AND LOCATIONS:
Locations (1):
- Plasma Physics Laboratory, National Institute of Nuclear Research, Ocoyoacac, State of Mexico, Mexico

IPD SHARING:
Plan to Share IPD: No